CLINICAL TRIAL: NCT06610032
Title: The Comparison O the Efficacy of Mesotherapy and Intra-articular Steroid Injection in Patients with Chronic Shoulder Pain
Brief Title: The Effect of Mesotherapy and Intra-articular Steroid Injection in Shoulder Pain
Acronym: Mesotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ecem Pelin Kaymaz, Medical Doctor of Physical Medicine and Rehabilitation, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMU-GETAT-EK 05/27.03.2024
Record Dates: First submitted 2024-08-26; First posted 2024-09-24 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Chronic Shoulder Pain
Keywords: Shoulder; Mesotherapy; Pain; Steroid Injection
MeSH Terms: conditions — Pain | interventions — Mesotherapy; Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mesotherapy (Active Comparator): A total of 3 sessions of mesotherapy will be applied to the shoulder area, 7 days apart.
  Interventions: Procedure: Mesotherapy
- Steroid (Active Comparator): A single-session intra-articular 20 mg triamcinolone hexacetonide injection will be administered.
  Interventions: Procedure: Intra-articular steroid injection

INTERVENTIONS:
Procedure: Mesotherapy — A total of 3 sessions of mesotherapy will be applied to the shoulder area of the patients, 7 days apart in group 1.
  Other Names: Intra-articular steroid injection
  Arms: Mesotherapy
Procedure: Intra-articular steroid injection — Single session intra-articular 20 mg triamcinolone hexacetonide injection will be applied for patients in group 2.
  Other Names: Mesotherapy
  Arms: Steroid

SUMMARY:
Patients with chronic shoulder pain will be divided randomly into mesotherapy and intra-articular steroid injection groups. Pain severity, range of motion and functional impairment will evaluated before treatment, 30 minutes and 4 weeks after the injections.

DETAILED DESCRIPTION:
The study will include 84 patients aged 18-75 who applied to physical medicine and rehabilitation out-patient clinic with chronic shoulder pain between May and July 2024. Patients will be randomly divided into two groups: a mesotherapy group and steroid injection group, using the closed-envelope method. In the first group, a total of 3 sessions of mesotherapy are applied to the shoulder areas of the patients, 7 days apart. A single-session intra-articular 20 mg triamcinolone hexacetonide injection will be administered for patients in group 2. Pain severity, range of motion and functional impairment will evaluated before treatment, 30 minutes and 4 weeks after the injections.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75
2. Having shoulder pain for 6 months
3. VAS (Visual Analog Scale) > 4
4. Patients who can receive verbal instructions and do not have cognitive deficits

Exclusion Criteria:

1. Physical therapy applied to the shoulder area in the last 3 months
2. Having had a shoulder joint injection in the last 3 months
3. History of previous upper extremity surgery
4. History of drug allergy
5. Use of anticoagulant drugs (warfarin, low molecular weight heparin), patients with coagulation disorder
6. History of malignancy
7. Psychiatric illness
8. A rheumatological diagnosis such as Polymyalgia Rheumatica, Rheumatoid Arthritis, Ankylosing Spondylitis
9. Kidney failure
10. Liver disease
11. Heart failure
12. Pregnancy
13. Presence of infection, wound, allergy, burn-like lesions in the application area

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
VAS (Visual Analouge Scale) | Patients will be evaluated before treatment, 30 minutes and 4 weeks after the injections.
  Pain Severity evaluation ((0 (no pain)-10 (unbearable pain))
Shoulder Disability Questionnaire' (OSS) form | Patients will be evaluated before treatment, 30 minutes and 4 weeks after the injections.
  Functional Disability evaluation (0-100)
Goniometric shoulder range of motion | Patients will be evaluated before treatment, 30 minutes and 4 weeks after the injections.
  shoulder range of motion evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University Haydarpasa Numune Research and Training Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mammucari M, Gatti A, Maggiori S, Sabato AF. Role of mesotherapy in musculoskeletal pain: opinions from the italian society of mesotherapy. Evid Based Complement Alternat Med. 2012;2012:436959. doi: 10.1155/2012/436959. Epub 2012 May 13. PMID 22654954
- [Background] Faetani L, Ghizzoni D, Ammendolia A, Costantino C. Safety and efficacy of mesotherapy in musculoskeletal disorders: A systematic review of randomized controlled trials with meta-analysis. J Rehabil Med. 2021 Apr 27;53(4):jrm00182. doi: 10.2340/16501977-2817. PMID 33764479